CLINICAL TRIAL: NCT05489744
Title: In Vivo Absorption, Metabolism, Excretion (AME) Clinical Study of [14C]Afuresertib in Healthy Chinese Male Adults - Human Mass Balance and Biotransformation Study of [14C]Afuresertib
Brief Title: Human Mass Balance and Biotransformation Study of [14C]Afuresertib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laekna Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LAE002CN1001
Record Dates: First submitted 2022-07-12; First posted 2022-08-05 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteer
Keywords: Mass balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 125 mg [14C]Afuresertib (Experimental): 125 mg/150 µCi [14C]Afuresertib (125 mg of Afuresertib containing 150 µCi of [14C]Afuresertib)
  Interventions: Drug: [14C]Afuresertib

INTERVENTIONS:
Drug: [14C]Afuresertib — Suspension containing approximately 125 mg of Afuresertib (containing 150 µCi of [14C]Afuresertib) is administered orally on an empty stomach, with approximately 240 mL of water for suspending and drug taking.
  Other Names: [14C]LAE002

SUMMARY:
This study adopts a single-center, single-dose, non-randomized, open-label design with a proposed enrollment of 6-10 healthy male subjects. After a single oral dose of approximately 125 mg/150 µCi [14C]Afuresertib tablets, blood, urine and fecal specimens are collected from each subject at defined time points/periods during the trial, and PK parameters, recovery, and excretion routes of [14C]Afuresertib in plasma are calculated by measuring the total radioactivity. The main metabolic and elimination pathways and characteristics of Afuresertib in human, as well as circulating metabolites with close to or higher than 10% of plasma total radioactivity exposure, are also identified by plasma, urine, and fecal radioactive metabolite profiles and major metabolite structure.

DETAILED DESCRIPTION:
This study includes two stages:

Stage I: The subjects are subject to the screening examination from D-7 to D-2. Two healthy adult male subjects selected from those who pass the examination are admitted to the clinical research center after qualification against the inclusion and exclusion criteria on D-2, and receive the baseline examination on D-1. After admission, they are trained on medication, urine and feces collection and other procedures to ensure that they can perform related operations in accordance with the protocol and operating manual for biospecimen analysis for mass balance and biotransformation study. Random urine and feces specimens (-24 h to 0 h) are collected on D-1 and the subjects are deprived of food for at least 10 h and water for 1 h before dosing. On the morning of the first day of the study, blood specimens are collected within 1 h before dosing, and the investigational product is taken orally on an empty stomach with 240 mL of warm water. The subjects are deprived of food for 4 h and water for 1 h after dosing. All urine and feces specimens excreted within the specified time intervals of 0-504 h and blood specimens sampled at specified time points before and within 0-504 h after dosing are collected. Phased testing is adopted in this study to determine whether specimen collection may be terminated in advance or the collection time needs to be prolonged based on the test results. If the specimen collection time exceeds 504 h, the collection should be extended at an interval of 24 h (urine, feces) or an integer multiple interval of 24 h (plasma) until the criteria for termination of specimen collection specified in the protocol are met. Meanwhile, the safety monitoring is continued until the completion date of the specimen collection.

Stage II: According to the results of the Stage I study, the necessarily for plan adjustment (dosing regimen, biospecimen collection, etc.) is evaluated, and another 4-8 subjects will be selected if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male adults;
2. Aged 18-45 years (inclusive);
3. BMI: 19-26 kg/m2 (inclusive); body weight ≥ 50 kg;
4. Willing to sign the Informed Consent Form (ICF);
5. Capable of communicating well with investigators and completing the entire study as required.

Exclusion Criteria:

1. Abnormal and clinically significant results of physical examination, vital signs, laboratory tests (routine hematology, blood biochemistry, coagulation function, routine urinalysis, fecal occult blood, thyroid function), 12-lead ECG, chest X-ray, and abdominal B-mode ultrasound (liver, gallbladder, pancreas, spleen, kidney);
2. Resting QT interval corrected with Fridericia's formula (QTcF) ≥ 450 ms shown on the 12-lead ECG;
3. Positive for hepatitis B surface antigen or E antigen, IgG antibody against hepatitis C virus (Anti-HCV IgG), antihuman immunodeficiency virus antigen/antibody (HIV-Ag/Ab) Combo Assay, and treponema pallidum antibody;
4. Clinically significant CRP abnormality in SaRS-CoV-2 infection screening or positive for SARS-CoV-2 nucleic acid test;
5. Use of any drug that inhibits or induces liver drug-metabolizing enzymes within 30 d before screening (see Appendix 1 for details);
6. Use of any prescription drugs, over-the-counter drugs, Chinese herbal medicines or food supplements, such as vitamins and calcium supplements, within 14 d before screening;
7. History of diabetes mellitus and/or pancreatitis;
8. History of any serious disease or condition that may affect the study results in the opinion of the investigators, including but not limited to disorders of the circulatory system, respiratory system, endocrine system, nervous system, digestive system, urinary system, or blood, immune, mentality, or metabolism diseases;
9. History of structural heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, torsades de pointes, ventricular tachycardia, atrioventricular block, long QT syndrome (LQTS), symptoms or family history of LQTS (indicated by genetic evidence or sudden death of close relatives due to cardiac causes at a young age);
10. Reception of major surgery (included but not limited to any surgery with significant risk of bleeding, prolonged general anesthesia, or significant traumatic injury, or incisional biopsy) within 6 months before the screening period, unhealed surgical wounds;
11. Allergic constitution, history of allergy to two or more substances; possibly allergic to the investigational product or its excipients as judged by the investigator;
12. Hemorrhoids or perianal disease with regular/ongoing hematochezia, irritable bowel syndrome, inflammatory bowel disease.
13. Habitual constipation or diarrhea;
14. Alcoholism or regular alcohol consumption within 6 months before screening period, that is, drinking volume > 14 U of alcohol per week (1 U = 360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine); breath alcohol test result > 0 mg/100 mL during the screening period;
15. Consumption of more than 5 cigarettes per day or habitual use of nicotine-containing products within 3 months before the screening period, and unable to abstain during the study;
16. Abuse of drugs or use of soft drugs (e.g., marijuana) 3 months before the screening period or use of hard drugs (e.g., cocaine, amphetamine, phencyclidine, etc.) 1 year before the screening period; or positive for urine drug test during the screening period;
17. Habitual consumption of grapefruit juice or excessive tea, coffee and/or caffeinated beverages, and unable to abstain during the study;
18. Long-term exposure to radioactivity, significant radioactive exposure (≥ 2 chest/abdomen CTs, or ≥ 3 other types of X-ray examinations) or participation in radiolabeled drug trials within 1 year prior to the study;
19. History of needle or blood sickness, difficulty in collecting blood, or intolerance of venipuncture blood collection;
20. Participation in any other clinical trial (including drug and device) within 3 months before the screening period;
21. Vaccination within 1 month before the screening period or scheduled vaccination during the study;
22. Scheduled for fathering or sperm donation during the study and within 1 year after the study; unwilling to take strict contraceptive measures during the study and within 1 year after the study (see Appendix 3 for details);
23. Blood loss or blood donation ≥ 400 mL within 3 months before the screening period, or blood transfusion within 1 month;
24. Any factors that render the subjects unsuitable for participating in this study (determined by the investigators).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-08-06 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Quantitatively analyze total radioactivity in the excreta. | 0-504 hours after IP taken. Phased testing is adopted in this study to determine whether specimen collection may be terminated in advance or the collection time needs to be prolonged based on the test results.
  Quantitatively analyze total radioactivity in the excreta of healthy male subjects after oral administration of [14C]Afuresertib to calculate the excretion of radioactivity in human body and confirm the main excretion route of the drug.
Pharmacokinetics (PK) analysis of radioactivity in plasma will be measured. | 0-504 hours after IP taken. Phased testing is adopted in this study to determine whether specimen collection may be terminated in advance or the collection time needs to be prolonged based on the test results.
  The total radioactivity in collected plasma and urine specimens is determined by a liquid scintillation counter.
  The collected whole blood and feces homogenate specimens are combusted by an oxidation combustor, and the total radioactivity is measured and calculated by a liquid scintillation counter.
Identify the main biotransformation pathways and the major metabolites by HPLC-MS/MS. | 0-504 hours after IP taken. Phased testing is adopted in this study to determine whether specimen collection may be terminated in advance or the collection time needs to be prolonged based on the test results.
  Each mixed specimen is processed by appropriate methods, and followed by the combination of HPLC and on-line or off-line isotope detector to obtain radioisotope metabolite profile.
  The major metabolites in plasma, urine and feces specimens are identified by HPLC-MS/MS.
  Cumulative recovery of total radioactivity in urine and/or feces will be measured by HPLC-MS/MS.
Quantitatively analyze the concentration of Afuresertib and its metabolites by the validated HPLC-MS/MS. | 0-504 hours after IP taken. Phased testing is adopted in this study to determine whether specimen collection may be terminated in advance or the collection time needs to be prolonged based on the test results.
  Quantitatively analyze the concentration of Afuresertib and its metabolites (if applicable) in plasma using a validated HPLC-MS/MS method to obtain the PK parameters in plasma.
  Percentage of each metabolite in urine and feces to the dose (%dose) or percentage of circulating metabolites in plasma to total exposure AUC (% AUC).

SECONDARY OUTCOMES:
Safety and tolerability of Afuresertib as measured by adverse events (AEs) . | During the screening period, at Day-2, Day-1, before dosing (within 1 hour before dosing) and at 4, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408, 432, 456, 480, and 504 hours after dosing.
  The cases of AEs, number of subjects and incidence are calculated, and listed by system organ class (SOC) and preferred term (PT). A detailed list of various AEs is also made. The severity of AEs and SAEs and the relationship with the investigational product are summarized separately.

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China